CLINICAL TRIAL: NCT05236062
Title: Impact of Exercise on the Complications of Corticosteroids in Patients With Graft-Versus-Host Disease Following Allogeneic Stem Cell Transplantation: the RESTART Trial
Brief Title: Impact of Exercise on the Complications of Corticosteroids in Patients With GVHD: the RESTART Trial
Acronym: RESTART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-618
Record Dates: First submitted 2022-01-19; First posted 2022-02-11 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Graft Vs Host Disease; Acute-graft-versus-host Disease; Chronic Graft-versus-host-disease
Keywords: Graft Vs Host Disease; Acute-graft-versus-host Disease; Chronic Graft-versus-host-disease; Corticosteroids; Allogeneic stem cell transplant
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Home-based, virtually supervised via Zoom, 3x weekly for 12-weeks aerobic and resistance exercise program
  Participants will also undergo four testing visits across 6-month period. Tests will include four blood draws and three body composition scans via a dual-energy x-ray absorptiometry (DXA).
  Interventions: Behavioral: Exercise
- Attention control Group (Experimental): Home-based, 12-week stretching program only with participants asked not to change their activity behavior.
  Participants will also undergo four testing visits across 6-month period. Tests will include four blood draws and three body composition scans via a dual-energy x-ray absorptiometry (DXA).
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Exercise — aerobic and resistance exercise
  Arms: Exercise Group
Behavioral: Attention control — stretching
  Arms: Attention control Group

SUMMARY:
This study is about determining if an aerobic and resistance exercise intervention is feasible in patients diagnosed with acute or chronic GVHD (Graft-Versus-Host Disease) after having an allogeneic stem cell transplant.

The names of the study interventions involved in this study are:

* Aerobic and resistance exercise (A+R) - Home-based aerobic and resistance exercise program
* Attention control (AC) - Home-based stretching program

DETAILED DESCRIPTION:
This research study is a feasibility study, which is the first-time investigators are examining an aerobic and resistance exercise (A+R) in patients diagnosed with acute or chronic GVHD after having an allogeneic stem cell transplant and if participating in a specific exercise program can improve glycemic control, body composition, physical fitness and function, and patient-reported outcomes.

This study consists of participants randomly assigned in 2(A+R):1(AC) ratio to one of two groups:

* Aerobic and resistance exercise (A+R), or
* Attention control (AC)

The A+R group will be asked to perform aerobic exercise, which can improve cardiovascular (heart) and lung function, and resistance exercise (e.g., dumbbell lifting), to help build muscle mass and strength. The AC group will be asked to perform stretching only and not to change their activity behavior.

All participants will also undergo four testing visits involving four blood draws and three body composition scans via a dual-energy x-ray absorptiometry (DXA).

Participants will be in this research study for 6 months.

It is expected that about 36 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old; children under the age of 18 will be excluded due to rarity of disease
* Newly diagnosed with acute or chronic GVHD, starting corticosteroids at a dose of 1 mg/kg or greater for the first time since transplant
* Received allogeneic stem cell transplant (any conditioning, any donor) at Dana-Farber Cancer Institute
* Physician's clearance to participate in moderate-vigorous intensity exercise
* Speak English
* Currently participate in less than 60 minutes of structured exercise/week
* Willing to travel to Dana-Farber Cancer Institute for necessary data collection
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Have a plan for hospital admission within the next 13 weeks at the time of recruitment
* If patients are not enrolled within 7 days after initial steroid treatment, they will be ineligible
* Pre-existing musculoskeletal or cardiorespiratory conditions
* Patients should not have any uncontrolled illness including ongoing or active infection, uncontrolled diabetes, hypertension, or thyroid disease
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* Patients with other active malignancies
* Participate in more than 60 minutes of structured exercise/week
* Unable to travel to Dana-Farber Cancer Institute for necessary data collection
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completing the exercise intervention sessions | 12 weeks
  The primary outcome is feasibility and will be assessed by the proportion of patients completing the exercise intervention sessions with >70% completion considered feasible.

SECONDARY OUTCOMES:
Glycemic control level | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Glycemic control level change will be measured by Homeostasis Model Assessment (HOMA). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Body Composition | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Body Composition Index change will be measured by Dual Energy X-Ray Absorptiometry (DEXA). Differences in lean mass, fat mass, and body fat % between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Cardiopulmonary Fitness | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Cardiopulmonary fitness will be measured by a submaximal graded exercise cycling test. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical function - Margaria Stair Climb | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Functional power will be measured using the Margaria Stair Climb test. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical Fitness | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Physical Fitness will be measured by the short physical performance battery (SPPB). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical Function - Handgrip Strength | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Handgrip strength will be measured by a hand-held dynamometer. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical Function - Timed Up and Go | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Physical function will be assessed with the timed-up-and-go (TUG) test. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical Function - 6 minute walk test | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Physical function will be assessed with the 6 minute walk test (6MWT). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Muscular Strength | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Muscular strength will be assessed with a 10 repetition maximum test. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Patient reported outcomes - Fatigue | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Fatigue will be measured by the PROMIS cancer fatigue short form. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Patient reported outcomes - Function | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Function will be measured by the Vulnerable Elders Survey (VES). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Patient reported outcomes - Quality of Life | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Quality of life will be assessed by the functional assessment of cancer therapy - bone marrow transplant (FACT-BMT). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Patient reported outcomes - Anxiety and Depression | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Anxiety and depression will be assessed by the Hospital Anxiety and Depression Scale (HADS). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Patient reported outcomes - Sleep | Evaluated at week 1 at baseline and week 7 on treatment, and at week 13 post-treatment also at week 25 follow-up
  Sleep will be assessed by the Pittsburg sleep quality index (PSQI). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu